CLINICAL TRIAL: NCT05547685
Title: Harmonic Generation Microscopy Observation of Intradermal Injection Nerve Fibers by Methylene Blue Intra-vital Staining
Brief Title: Methylene Blue Intra-vital Nerve Staining
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201904083MINA
Record Dates: First submitted 2020-08-30; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-01

CONDITIONS: Neurologic Findings
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methylene blue intradermal injection (Experimental): Methylene blue intradermal injection
  Interventions: Diagnostic Test: Methylene blue intradermal injection

INTERVENTIONS:
Diagnostic Test: Methylene blue intradermal injection — Methylene blue intradermal injection

SUMMARY:
In previous studies, we know methylene blue (MB) stains nerves, and oxidized MB has near-infrared (NIR) fluorescence for fluorescent observation. In this trial we using MB on human skin and combining MB and third-harmonic generation imaging (THG) to label cutaneous nerve fibers.

DETAILED DESCRIPTION:
Intravital images were obtained before injection and then taken at 0.5, 1, 1.5, 2, 2.5, and 3 h after intradermal 0.03% (0.3 mg/mL, 1500μM) MB (10mg/mL "Astar") injection using a 0.5-mL 29-gauge insulin syringe needle (Becton, Dickinson and Company, USA). The participant lay down and the skin was imaged 10 cm above the ankle in the lower leg and above the wrist in the middle forearm; three sites in each limb were randomly selected for each time point. SHG or THG captured MB signals with two-photon excitation microscope at the Molecular Biomedical Imaging Research Center of National Taiwan University.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers

Exclusion Criteria:

* used serotonin agonist medication

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-10-17 (Estimated); Study Completion 2022-10-17 (Estimated)

PRIMARY OUTCOMES:
intravital staining | 12 months
  injected 10 μL of 0.03% methylene blue intradermally then calculate nerve fiber image

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hosipital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided